CLINICAL TRIAL: NCT00356135
Title: A Pharmacodynamic Comparison of Prasugrel (LY640315) Versus Clopidogrel in Subjects With Acute Coronary Syndrome Who Are Receiving Clopidogrel
Brief Title: Effect of Prasugrel on Platelets After One Week in Patients Already Taking Clopidogrel After a Cardiac Event
Acronym: SWAP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Daiichi Sankyo (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 10631; H7T-MC-TABM (Other: Eli Lilly and Company)
Record Dates: First submitted 2006-07-21; First posted 2006-07-25 (Estimated); Results first posted 2010-03-09 (Estimated); Last update posted 2010-11-03 (Estimated); Status verified 2010-10

CONDITIONS: Coronary Arteriosclerosis; Acute Coronary Syndrome
MeSH Terms: conditions — Coronary Artery Disease; Acute Coronary Syndrome | interventions — Prasugrel Hydrochloride; Clopidogrel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- Prasugrel 10/10 mg (Experimental): Open label (lead-in) dose of clopidogrel 75 milligram (mg) for 10 to 14 days. Upon completion, assignment to a single loading dose of prasugrel 10 mg and placebo, followed by maintenance dose of prasugrel 10 mg taken for 13 to 15 days.
  Interventions: Drug: prasugrel 10 mg; Drug: clopidogrel; Drug: prasugrel placebo; Drug: clopidogrel placebo
- Clopidogrel 75/75 mg (Experimental): Open label (lead-in) dose of clopidogrel 75 mg for 10 to 14 days. Upon completion, assignment to a single loading dose of clopidogrel 75 mg and placebo, followed by maintenance dose of clopidogrel 75 mg taken for 13 to 15 days.
  Interventions: Drug: clopidogrel; Drug: prasugrel placebo
- Prasugrel 60/10 mg (Experimental): Open label (lead-in) dose of clopidogrel 75 mg for 10 to 14 days. Upon completion, assignment to a single loading dose of prasugrel 60 mg and placebo followed by maintenance dose of prasugrel 10 mg taken for 13 to 15 days.
  Interventions: Drug: prasugrel 10 mg; Drug: clopidogrel; Drug: prasugrel 60 mg; Drug: clopidogrel placebo

INTERVENTIONS:
Drug: prasugrel 10 mg — 10 mg tablet taken orally
  Other Names: LY640315; Effient; Efient
  Arms: Prasugrel 10/10 mg; Prasugrel 60/10 mg
Drug: clopidogrel — 75 mg tablet taken orally
  Other Names: Plavix; Clopilet; Clavix
Drug: prasugrel placebo — oral, as blinding mechanism.
  Arms: Clopidogrel 75/75 mg; Prasugrel 10/10 mg
Drug: prasugrel 60 mg — 60 mg (six 10-mg tablets) taken orally
  Other Names: LY640315; Effient; Efient
  Arms: Prasugrel 60/10 mg
Drug: clopidogrel placebo — oral, as blinding mechanism
  Arms: Prasugrel 10/10 mg; Prasugrel 60/10 mg

SUMMARY:
This study will compare the effect of a prasugrel 10-mg maintenance dose with a clopidogrel 75-mg maintenance dose on platelet activity, approximately 1 week after the first dose of study drug, in subjects who have been taking clopidogrel 75 mg daily following a percutaneous coronary intervention (PCI) with placement of a stent, performed to treat acute coronary syndrome (ACS).

ELIGIBILITY:
Inclusion Criteria:

* Present with a recent history of an ACS event based on the disease diagnostic criteria between 30 and 330 days prior to enrollment, and who state that they are supposed to be taking daily aspirin and maintenance dose 75-mg clopidogrel.
* Are of a legal age (and at least 18 years of age but less than 75 years of age) and competent mental condition to provide written informed consent before entering the study.

Exclusion Criteria:

* Left main coronary artery stent or left anterior descending (LAD) bifurcation stent.
* Have any form of coronary revascularization (percutaneous coronary intervention [PCI] or coronary artery bypass grafting [CABG]) planned to occur during the study (from signing consent through the final visit).
* Have undergone CABG or PCI within 30 days of entry into the study.
* Receiving or will receive oral anticoagulation or other antiplatelet therapy (other than aspirin and clopidogrel) that cannot be safely discontinued for the duration of the study.
* Receiving daily treatment with nonsteroidal anti-inflammatory drugs (NSAIDs) that cannot be discontinued or are anticipated to require daily treatment with NSAIDs during the study.
* Have any of the following: history of ischemic or hemorrhagic stroke intracranial neoplasm, arteriovenous malformation, or aneurysm history of transient ischemic attack (TIA), have a body weight less than 60 kilograms (kg).

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2006-07; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 317-615-4559 Mon - Fri 9 am - 5 pm Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (9):
- United States (9):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Jacksonville, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Baltimore, Maryland
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Worcester, Massachusetts
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Ann Arbor, Michigan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Cincinnati, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Columbus, Ohio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Oklahoma City, Oklahoma
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Rapid City, South Dakota
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Monday-Friday from 9:00 AM to 5:00 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician, Houston, Texas

REFERENCES:
- [Result] Angiolillo DJ, Saucedo JF, Deraad R, Frelinger AL, Gurbel PA, Costigan TM, Jakubowski JA, Ojeh CK, Effron MB; SWAP Investigators. Increased platelet inhibition after switching from maintenance clopidogrel to prasugrel in patients with acute coronary syndromes: results of the SWAP (SWitching Anti Platelet) study. J Am Coll Cardiol. 2010 Sep 21;56(13):1017-23. doi: 10.1016/j.jacc.2010.02.072. PMID 20846599
- [Derived] Saucedo JF, Angiolillo DJ, DeRaad R, Frelinger AL 3rd, Gurbel PA, Costigan TM, Jakubowski JA, Ojeh CK, Duvvuru S, Effron MB; SWAP Investigators. Decrease in high on-treatment platelet reactivity (HPR) prevalence on switching from clopidogrel to prasugrel: insights from the switching anti-platelet (SWAP) study. Thromb Haemost. 2013 Feb;109(2):347-55. doi: 10.1160/TH12-06-0378. Epub 2012 Dec 6. PMID 23223867

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 30-330 days after acute coronary syndrome event, patients participated in 2 week open-label clopidogrel phase. Patients were then randomized to either 22-26 hour loading doses of: 60-mg prasugrel, 10-mg prasugrel, or 75-mg clopidogrel, then continued 2-week maintenance phase of 10-mg prasugrel, 10-mg prasugrel, or 75-mg clopidogrel, respectively.
Groups:
- Prasgurel 10/10 mg: Open label dose of clopidogrel 75 milligram (mg) for 10 to 14 days. Upon completion, randomized to a single loading dose of prasugrel 10 mg and placebo, followed by maintenance dose of prasugrel 10 mg taken for 13 to 15 days.
- Clopidogrel 75/75 mg: Open label dose of clopidogrel 75 mg for 10 to 14 days. Upon completion, randomized to a single loading dose of clopidogrel 75 mg and placebo, followed by maintenance dose of clopidogrel 75 mg taken for 13 to 15 days.
- Prasugrel 60/10 mg: Open label dose of clopidogrel 75 mg for 10 to 14 days. Upon completion, randomized to a single loading dose of prasugrel 60 mg and placebo followed by maintenance dose of prasugrel 10 mg taken for 13 to 15 days.
Period: Overall Study
Arm/Group | Prasgurel 10/10 mg | Clopidogrel 75/75 mg | Prasugrel 60/10 mg
Started | 47 | 48 | 44
Completed | 43 | 46 | 39
Not Completed | 4 | 2 | 5
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Physician Decision | 1 | 1 | 1
Not completed — Subject non-compliance | 1 | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Prasugrel 10/10 mg: Open label dose of clopidogrel 75 milligram (mg) for 10 to 14 days. Upon completion, randomization to a single loading dose of prasugrel 10 mg and placebo, followed by maintenance dose of prasugrel 10 mg taken for 13 to 15 days.
- Clopidogrel 75/75 mg: Open label dose of clopidogrel 75 mg for 10 to 14 days. Upon completion, randomization to a single loading dose of clopidogrel 75 mg and placebo, followed by maintenance dose of clopidogrel 75 mg taken for 13 to 15 days.
- Total: Total of all reporting groups
Arm/Group | Prasugrel 10/10 mg | Clopidogrel 75/75 mg | Prasugrel 60/10 mg | Total
Number analyzed (Participants) | 47 | 48 | 44 | 139
Age Continuous [Mean (Standard Deviation); unit: years] | 57.6 (8.18) | 56.9 (8.93) | 58.7 (9.16) | 57.7 (8.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 18 | 15 | 45
  Male | 35 | 30 | 29 | 94
Race/Ethnicity, Customized [Number; unit: participants] — breakdown of participants by race/ethnicity
  participants
    Caucasian | 39 | 30 | 37 | 106
    African | 7 | 13 | 6 | 26
    Asian | 0 | 0 | 0 | 0
    Other | 1 | 5 | 1 | 7
Region of Enrollment [Number; unit: participants]
  United States | 47 | 48 | 44 | 139

OUTCOME MEASURES:

1. Primary Outcome: Maximum Platelet Aggregation (MPA) to 20 Micromolar (uM) Adenosine Diphosphase (ADP)
Description: Maximum platelet aggregation (MPA) to 20 micromolar adenosine diphosphase (ADP) as measured with light transmittance aggregometry (LTA).
Time Frame: 1 week after first dose of randomized study drug
Population: The primary analysis population was the pharmacodynamic (PD) population which included all randomized participants who had blood draws for MPA at 1 week after randomization who met compliance criteria, and who had last dose of study drug the day prior to the blood draw for MPA.
Measure: Least Squares Mean (Standard Error); unit: percent maximum platelet aggregation (%)
Groups:
- Prasugrel 60/10 mg: Open label dose of clopidogrel 75 mg for 10 to 14 days. Upon completion, randomization to a single loading dose of prasugrel 60 mg and placebo followed by maintenance dose of prasugrel 10 mg taken for 13 to 15 days.
Arm/Group | Prasugrel 10/10 mg | Clopidogrel 75/75 mg | Prasugrel 60/10 mg
Number analyzed (Participants) | 34 | 31 | 30
percent maximum platelet aggregation (%) | 41.1 (1.99) | 55.0 (2.09) | 41.0 (2.00)
Statistical Analysis 1: Comparison: Prasugrel 10/10 mg vs Clopidogrel 75/75 mg; Test type: Superiority or Other; p < 0.0001, ANOVA; Treatment and study sites are fixed effects and MPA right before the randomization treatment period is a covariate in the model; Mean Difference (Final Values) = -13.91, 95% CI [-19.10 to -8.73] — Mean Difference is for Prasugrel 10/10 mg arm minus Clopidogrel 75/75 mg arm
Statistical Analysis 2: Comparison: Clopidogrel 75/75 mg vs Prasugrel 60/10 mg; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -13.98, 95% CI [-19.26 to -8.71]

2. Secondary Outcome: Maximum Platelet Aggregation (MPA) (to 5 and 20 uM ADP) at 2 Hours, 24 Hours, 1 Week and 2 Weeks
Description: Maximum platelet aggregation (MPA) to 5 and 20 micromolar adenosine diphosphase (ADP) as measured with light transmittance aggregometry (LTA).
Time Frame: 2 hours, 24 hours, 1 week, 2 weeks after first dose of randomized study drug
Population: Pharmacodynamic Population, which included all randomized participants who had blood draws for MPA, who met compliance criteria, and who had last dose of study drug the day prior to the blood draw for MPA.
Measure: Mean (Standard Deviation); unit: percent maximum platelet aggregation (%)
Arm/Group | Prasugrel 10/10 mg | Clopidogrel 75/75 mg | Prasugrel 60/10 mg
Number analyzed (Participants) | 36 | 33 | 31
percent maximum platelet aggregation (%)
  2 Hour (20 uM ADP) | 49.46 (21.243) [-8.22 to 3.35] | 48.07 (17.728) [-29.30 to -17.51] | 26.65 (10.875)
  24 Hour (20 uM ADP) | 52.29 (16.511) [-8.82 to 0.32] | 53.80 (14.504) [-33.20 to -23.94] | 27.36 (10.812)
  1 Week (20 uM ADP) | 42.95 (14.963) [-19.96 to -9.65] | 53.80 (14.878) [-19.87 to -9.32] | 40.64 (10.182)
  2 Week (20 uM ADP) | 40.84 (13.359) [-20.30 to -9.22] | 52.25 (16.856) [-20.59 to -9.22] | 38.61 (13.373)
  2 Hour (5 uM ADP) | 37.87 (16.547) [-5.85 to 3.14] | 37.25 (12.579) [-21.55 to -12.37] | 19.97 (11.263)
  24 Hour (5 uM ADP) | 38.84 (14.841) [-8.58 to 0.42] | 40.88 (14.540) [-24.81 to -15.64] | 20.94 (11.476)
  1 Week (5 uM ADP) | 32.44 (11.739) [-17.21 to -7.50] | 41.94 (14.436) [-15.79 to -5.79] | 31.45 (11.446)
  2 Week (5 uM ADP) | 30.18 (11.444) [-17.41 to -7.72] | 41.05 (13.570) [-16.80 to -6.82] | 28.64 (13.534)
Statistical Analysis 1: Comparison: Prasugrel 10/10 mg vs Clopidogrel 75/75 mg; Test type: Superiority or Other; p = 0.4055, Repeated Measures Analysis — P-value for 2 Hour (20 uM ADP). Mixed model with actual value at each timepoint as dependent variable, baseline value as covariate, treatment, catagorical timepoint, and time by treatment interaction as fixed effects, and subject as random effect; Least Squares Mean Difference = -2.4, 95% CI 2-sided [-8.22 to 3.35] — Least Squares Mean Difference = Prasugrel 10/10 mg minus Clopidogrel 75/75 mg
Statistical Analysis 2: Comparison: Clopidogrel 75/75 mg vs Prasugrel 60/10 mg; Test type: Superiority or Other; p < 0.0001, Repeated Measures Analysis — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -23, 95% CI 2-sided [-29.30 to -17.51] — Least Squares Mean Difference = Prasugrel 60/10 mg minus Clopidogrel 75/75 mg
Statistical Analysis 3: Comparison: Prasugrel 10/10 mg vs Clopidogrel 75/75 mg; Test type: Superiority or Other; p = 0.0680, Repeated Measures Analysis — P-value for 24 Hour (20 uM ADP). Mixed model with actual value at each timepoint as dependent variable, baseline value as covariate, treatment, catagorical timepoint, and time by treatment interaction as fixed effects, and subject as random effect; Least Squares Mean Difference = -4.2, 95% CI 2-sided [-8.82 to 0.32] — Least Squares Mean Difference = Prasugrel 10/10 mg minus Clopidogrel 75/75 mg
Statistical Analysis 4: Comparison: Clopidogrel 75/75 mg vs Prasugrel 60/10 mg; Comparison of MPA to 20 uM ADP at 24 hours; Test type: Superiority or Other; p < 0.0001, Repeated Measures Analysis — [p-value comment as in outcome 2, analysis 3]; Least Squares Mean Difference = -29, 95% CI 2-sided [-33.20 to -23.94] — Least Squares Mean Difference = Prasugrel 60/10 mg minus Clopidogrel 75/75 mg
Statistical Analysis 5: Comparison: Prasugrel 10/10 mg vs Clopidogrel 75/75 mg; Test type: Superiority or Other; p < 0.0001, Repeated Measures Analysis — P-value for 1 Week (20 uM ADP). Mixed model with actual value at each timepoint as dependent variable, baseline value as covariate, treatment, catagorical timepoint, and time by treatment interaction as fixed effects, and subject as random effect; Least Squares Mean Difference = -15, 95% CI 2-sided [-19.96 to -9.65] — Least Squares Mean Difference = Prasugrel 10/10 mg minus Clopidogrel 75/75 mg
Statistical Analysis 6: Comparison: Clopidogrel 75/75 mg vs Prasugrel 60/10 mg; Test type: Superiority or Other; p < 0.0001, Repeated Measures Analysis — [p-value comment as in outcome 2, analysis 5]; Least Squares Mean Difference = -15, 95% CI 2-sided [-19.87 to -9.32] — Least Squares Mean Difference = Prasugrel 60/10 mg minus Clopidogrel 75/75 mg
Statistical Analysis 7: Comparison: Prasugrel 10/10 mg vs Clopidogrel 75/75 mg; Test type: Superiority or Other; p < 0.0001, Repeated Measures Analysis — P-value for 2 Week (20 uM ADP). Mixed model with actual value at each timepoint as dependent variable, baseline value as covariate, treatment, catagorical timepoint, and time by treatment interaction as fixed effects, and subject as random effect; Least Squares Mean Difference = -15, 95% CI 2-sided [-20.30 to -9.22] — Least Squares Mean Difference = Prasugrel 10/10 mg minus Clopidogrel 75/75 mg
Statistical Analysis 8: Comparison: Clopidogrel 75/75 mg vs Prasugrel 60/10 mg; Test type: Superiority or Other; p < 0.0001, Repeated Measures Analysis — [p-value comment as in outcome 2, analysis 7]; Least Squares Mean Difference = -15, 95% CI 2-sided [-20.59 to -9.22] — Least Squares Mean Difference = Prasugrel 60/10 mg minus Clopidogrel 75/75 mg
Statistical Analysis 9: Comparison: Prasugrel 10/10 mg vs Clopidogrel 75/75 mg; Test type: Superiority or Other; p = 0.5501, Repeated Measures Analysis — P-value for 2 Hour (5 uM ADP). Mixed model with actual value at each timepoint as dependent variable, baseline value as covariate, treatment, catagorical timepoint, and time by treatment interaction as fixed effects, and subject as random effect; Least Squares Mean Difference = -1.4, 95% CI 2-sided [-5.85 to 3.14] — Least Squares Mean Difference = Prasugrel 10/10 mg minus Clopidogrel 75/75 mg
Statistical Analysis 10: Comparison: Clopidogrel 75/75 mg vs Prasugrel 60/10 mg; Test type: Superiority or Other; p < 0.0001, Repeated Measures Analysis — [p-value comment as in outcome 2, analysis 9]; Least Squares Mean Difference = -17, 95% CI 2-sided [-21.55 to -12.37] — Least Squares Mean Difference = Prasugrel 60/10 mg minus Clopidogrel 75/75 mg
Statistical Analysis 11: Comparison: Prasugrel 10/10 mg vs Clopidogrel 75/75 mg; Test type: Superiority or Other; p = 0.0752, Repeated Measures Analysis — P-value for 24 Hour (5 uM ADP). Mixed model with actual value at each timepoint as dependent variable, baseline value as covariate, treatment, catagorical timepoint, and time by treatment interaction as fixed effects, and subject as random effect; Least Squares Mean Difference = -4.1, 95% CI 2-sided [-8.58 to 0.42] — Least Squares Mean Difference = Prasugrel 10/10 mg minus Clopidogrel 75/75 mg
Statistical Analysis 12: Comparison: Clopidogrel 75/75 mg vs Prasugrel 60/10 mg; Test type: Superiority or Other; p < 0.0001, Repeated Measures Analysis — [p-value comment as in outcome 2, analysis 11]; Least Squares Mean Difference = -20, 95% CI 2-sided [-24.81 to -15.64] — Least Squares Mean Difference = Prasugrel 60/10 mg minus Clopidogrel 75/75 mg
Statistical Analysis 13: Comparison: Prasugrel 10/10 mg vs Clopidogrel 75/75 mg; Test type: Superiority or Other; p < 0.0001, Repeated Measures Analysis — P-value for 1 Week (5 uM ADP). Mixed model with actual value at each timepoint as dependent variable, baseline value as covariate, treatment, catagorical timepoint, and time by treatment interaction as fixed effects, and subject as random effect; Least Squares Mean Difference = -12, 95% CI 2-sided [-17.21 to -7.50] — Least Squares Mean Difference = Prasugrel 10/10 mg minus Clopidogrel 75/75 mg
Statistical Analysis 14: Comparison: Clopidogrel 75/75 mg vs Prasugrel 60/10 mg; Test type: Superiority or Other; p < 0.0001, Repeated Measures Analysis — [p-value comment as in outcome 2, analysis 13]; Least Squares Mean Difference = -11, 95% CI 2-sided [-15.79 to -5.79] — Least Squares Mean Difference = Prasugrel 60/10 mg minus Clopidogrel 75/75 mg
Statistical Analysis 15: Comparison: Prasugrel 10/10 mg vs Clopidogrel 75/75 mg; Test type: Superiority or Other; p < 0.0001, Repeated Measures Analysis — P-value for 2 Week (5 uM ADP). Mixed model with actual value at each timepoint as dependent variable, baseline value as covariate, treatment, catagorical timepoint, and time by treatment interaction as fixed effects, and subject as random effect; Least Squares Mean Difference = -13, 95% CI 2-sided [-17.41 to -7.72] — Least Squares Mean Difference = Prasugrel 10/10 mg minus Clopidogrel 75/75 mg
Statistical Analysis 16: Comparison: Clopidogrel 75/75 mg vs Prasugrel 60/10 mg; Test type: Superiority or Other; p < 0.0001, Repeated Measures Analysis — [p-value comment as in outcome 2, analysis 15]; Least Squares Mean Difference = -12, 95% CI 2-sided [-16.80 to -6.82] — Least Squares Mean Difference = Prasugrel 60/10 mg minus Clopidogrel 75/75 mg

3. Secondary Outcome: Maximum Platelet Aggregation (MPA) to 20 uM ADP According to Clopidogrel Use at Time of Qualifying Acute Coronary Syndrome (ACS) Event
Description: Data provided are the MPA to 20 micromolar ADP while taking clopidogrel (measurement taken at end of the 14 day open label phase) grouped by subjects who were taking clopidogrel at the time of the qualifying ACS event compared with subjects who were not taking clopidogrel at the time of the qualifying ACS event.
Time Frame: End of 14 day open label
Population: Pharmacodynamic Population, which included all randomized participants who had blood draws for MPA, who met compliance criteria, and who had last dose of study drug the day prior to the blood draw for MPA. Grouped according to clopidogrel use at time of ACS event and no clopidogrel use at time of ACS event.
Measure: Mean (Standard Deviation); unit: percent maximum platelet aggregation (%)
Groups:
- Clopidogrel Use: Patients with clopidogrel use at the time of qualifying ACS event.
- No Clopidogrel Use: Patients with no clopidogrel use at the time of qualifying ACS event.
Arm/Group | Clopidogrel Use | No Clopidogrel Use
Number analyzed (Participants) | 20 | 75
percent maximum platelet aggregation (%) | 60.73 (18.729) | 55.53 (14.356)
Statistical Analysis 1: Comparison: Clopidogrel Use vs No Clopidogrel Use; The mean of MPA 20 uM ADP at the end of Clopidogrel open label of patients on chronic clopidogrel at the time of qualifying events was compared to the mean MPA of patients not using clopidogrel at this time; Test type: Superiority or Other; p = 0.1824, t-test, 2 sided
Statistical Analysis 2: Comparison: Clopidogrel Use vs No Clopidogrel Use; The variance of MPA 20 uM ADP at the end of Clopidogrel open label of patients on chronic clopidogrel at the time of qualifying events was compared to the variance of MPA for patients not using clopidogrel at this time; Test type: Superiority or Other; p = 0.1101, F-test

4. Secondary Outcome: Residual Platelet Aggregation (RPA) (to 5 and 20 uM ADP) at 2 Hours, 24 Hours, 1 Week and 2 Weeks
Description: Residual platelet aggregation after the addition 5 and 20 micromolar ADP as measured with light transmittance aggregometry (LTA).
Time Frame: 2 hours, 24 hours, 1 week, 2 weeks after first dose of randomized study drug
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent residual platelet aggregation
Arm/Group | Prasugrel 10/10 mg | Clopidogrel 75/75 mg | Prasugrel 60/10 mg
Number analyzed (Participants) | 36 | 33 | 31
percent residual platelet aggregation
  2 Hour (20 uM ADP) | 32.06 (24.462) [-9.50 to 3.37] | 28.21 (21.792) [-33.40 to -20.33] | 5.10 (7.814)
  24 Hour (20 uM ADP) | 32.97 (21.858) [-13.04 to -1.60] | 35.16 (19.379) [-39.99 to -28.42] | 4.70 (5.688)
  1 Week (20 uM ADP) | 22.92 (17.961) [-25.58 to -11.09] | 34.45 (21.752) [-27.09 to -12.26] | 17.94 (12.961)
  2 Week (20 uM ADP) | 18.89 (14.401) [-28.42 to -14.77] | 34.56 (19.515) [-29.61 to -15.63] | 15.17 (15.127)
  2 Hour (5 uM ADP) | 18.83 (17.574) [-3.11 to 6.38] | 14.84 (12.767) [-15.92 to -6.24] | 4.17 (4.878)
  24 Hour (5 uM ADP) | 19.18 (16.448) [-8.31 to 1.74] | 19.66 (14.672) [-20.98 to -10.75] | 4.45 (4.545)
  1 Week (5 uM ADP) | 11.11 (10.325) [-18.81 to -7.32] | 21.57 (18.829) [-17.91 to -6.09] | 9.94 (10.370)
  2 Week (5 uM ADP) | 10.03 (9.247) [-15.64 to -6.32] | 19.28 (14.824) [-14.67 to -5.09] | 9.43 (8.621)
Statistical Analysis 1: Comparison: Prasugrel 10/10 mg vs Clopidogrel 75/75 mg; Test type: Superiority or Other; p = 0.3466, Repeated Measures Analysis — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -3.1, 95% CI 2-sided [-9.50 to 3.37] — Least Squares Mean Difference = Prasugrel 10/10 mg minus Clopidogrel 75/75 mg
Statistical Analysis 2: Comparison: Clopidogrel 75/75 mg vs Prasugrel 60/10 mg; Test type: Superiority or Other; p < 0.0001, Repeated Measures Analysis — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -27, 95% CI 2-sided [-33.40 to -20.33] — Least Squares Mean Difference = Prasugrel 60/10 mg minus Clopidogrel 75/75 mg
Statistical Analysis 3: Comparison: Prasugrel 10/10 mg vs Clopidogrel 75/75 mg; Test type: Superiority or Other; p = 0.0127, Repeated Measures Analysis — [p-value comment as in outcome 2, analysis 3]; Least Squares Mean Difference = -7.3, 95% CI 2-sided [-13.04 to -1.60] — Least Squares Mean Difference = Prasugrel 10/10 mg minus Clopidogrel 75/75 mg
Statistical Analysis 4: Comparison: Clopidogrel 75/75 mg vs Prasugrel 60/10 mg; Test type: Superiority or Other; p < 0.0001, Repeated Measures Analysis — [p-value comment as in outcome 2, analysis 3]; Least Squares Mean Difference = -34, 95% CI 2-sided [-39.99 to -28.42] — Least Squares Mean Difference = Prasugrel 60/10 mg minus Clopidogrel 75/75 mg
Statistical Analysis 5: Comparison: Prasugrel 10/10 mg vs Clopidogrel 75/75 mg; Test type: Superiority or Other; p < 0.0001, Repeated Measures Analysis — [p-value comment as in outcome 2, analysis 5]; Least Squares Mean Difference = -18, 95% CI 2-sided [-25.58 to -11.09] — Least Squares Mean Difference = Prasugrel 10/10 mg minus Clopidogrel 75/75 mg
Statistical Analysis 6: Comparison: Clopidogrel 75/75 mg vs Prasugrel 60/10 mg; Test type: Superiority or Other; p < 0.0001, Repeated Measures Analysis — [p-value comment as in outcome 2, analysis 5]; Least Squares Mean Difference = -20, 95% CI 2-sided [-27.09 to -12.26] — Least Squares Mean Difference = Prasugrel 60/10 mg minus Clopidogrel 75/75 mg
Statistical Analysis 7: Comparison: Prasugrel 10/10 mg vs Clopidogrel 75/75 mg; Test type: Superiority or Other; p < 0.0001, Repeated Measures Analysis — [p-value comment as in outcome 2, analysis 7]; Least Squares Mean Difference = -22, 95% CI 2-sided [-28.42 to -14.77] — Least Squares Mean Difference = Prasugrel 10/10 mg minus Clopidogrel 75/75 mg
Statistical Analysis 8: Comparison: Clopidogrel 75/75 mg vs Prasugrel 60/10 mg; Test type: Superiority or Other; p < 0.0001, Repeated Measures Analysis — [p-value comment as in outcome 2, analysis 7]; Least Squares Mean Difference = -23, 95% CI 2-sided [-29.61 to -15.63] — Least Squares Mean Difference = Prasugrel 60/10 mg minus Clopidogrel 75/75 mg
Statistical Analysis 9: Comparison: Prasugrel 10/10 mg vs Clopidogrel 75/75 mg; Test type: Superiority or Other; p = 0.4954, Repeated Measures Analysis — [p-value comment as in outcome 2, analysis 9]; Least Squares Mean Difference = 1.6, 95% CI 2-sided [-3.11 to 6.38] — Least Squares Mean Difference = Prasugrel 10/10 mg minus Clopidogrel 75/75 mg
Statistical Analysis 10: Comparison: Clopidogrel 75/75 mg vs Prasugrel 60/10 mg; Test type: Superiority or Other; p < 0.0001, Repeated Measures Analysis — [p-value comment as in outcome 2, analysis 9]; Least Squares Mean Difference = -11, 95% CI 2-sided [-15.92 to -6.24] — Least Squares Mean Difference = Prasugrel 60/10 mg minus Clopidogrel 75/75 mg
Statistical Analysis 11: Comparison: Prasugrel 10/10 mg vs Clopidogrel 75/75 mg; Test type: Superiority or Other; p = 0.1971, Repeated Measures Analysis — [p-value comment as in outcome 2, analysis 11]; Least Squares Mean Difference = -3.3, 95% CI 2-sided [-8.31 to 1.74] — Least Squares Mean Difference = Prasugrel 10/10 mg minus Clopidogrel 75/75 mg
Statistical Analysis 12: Comparison: Clopidogrel 75/75 mg vs Prasugrel 60/10 mg; Test type: Superiority or Other; p < 0.0001, Repeated Measures Analysis — [p-value comment as in outcome 2, analysis 11]; Least Squares Mean Difference = -16, 95% CI 2-sided [-20.98 to -10.75] — Least Squares Mean Difference = Prasugrel 60/10 mg minus Clopidogrel 75/75 mg
Statistical Analysis 13: Comparison: Prasugrel 10/10 mg vs Clopidogrel 75/75 mg; Test type: Superiority or Other; p < 0.0001, Repeated Measures Analysis — [p-value comment as in outcome 2, analysis 13]; Least Squares Mean Difference = -13, 95% CI 2-sided [-18.81 to -7.32] — Least Squares Mean Difference = Prasugrel 10/10 mg minus Clopidogrel 75/75 mg
Statistical Analysis 14: Comparison: Clopidogrel 75/75 mg vs Prasugrel 60/10 mg; Test type: Superiority or Other; p = 0.0001, Repeated Measures Analysis — [p-value comment as in outcome 2, analysis 13]; Least Squares Mean Difference = -12, 95% CI 2-sided [-17.91 to -6.09] — Least Squares Mean Difference = Prasugrel 60/10 mg minus Clopidogrel 75/75 mg
Statistical Analysis 15: Comparison: Prasugrel 10/10 mg vs Clopidogrel 75/75 mg; Test type: Superiority or Other; p < 0.0001, Repeated Measures Analysis — [p-value comment as in outcome 2, analysis 15]; Least Squares Mean Difference = -11, 95% CI 2-sided [-15.64 to -6.32] — Least Squares Mean Difference = Prasugrel 10/10 mg minus Clopidogrel 75/75 mg
Statistical Analysis 16: Comparison: Clopidogrel 75/75 mg vs Prasugrel 60/10 mg; Test type: Superiority or Other; p < 0.0001, Repeated Measures Analysis — [p-value comment as in outcome 2, analysis 15]; Least Squares Mean Difference = -9.9, 95% CI 2-sided [-14.67 to -5.09] — Least Squares Mean Difference = Prasugrel 60/10 mg minus Clopidogrel 75/75 mg

5. Secondary Outcome: Correlation Coefficent of Verify Now™ P2Y12 Assay Values to Maximum Platelet Aggregation (MPA) and Residual Platelet Aggregation (RPA) to 20 uM ADP at 1 Week
Description: Correlation Coefficient comparing the Accumetrics VerifyNow™ P2Y12 device with light transmittance aggregometry (LTA) for monitoring platelet aggregation.
Time Frame: 1 week after randomized study drug
Population: as for outcome 2
Measure: Number; unit: correlation coefficient
Arm/Group | Prasugrel 10/10 mg | Clopidogrel 75/75 mg | Prasugrel 60/10 mg
Number analyzed (Participants) | 36 | 33 | 31
correlation coefficient
  MPA (20 uM ADP) at 1 week | 0.564 | 0.426 | 0.439
  RPA (20 uM ADP) at 1 week | 0.640 | 0.425 | 0.547
Statistical Analysis 1: Comparison: Prasugrel 10/10 mg; Test type: Superiority or Other; p = 0.0005, Pearson Correlation Coefficient — P-value for MPA (20 uM ADP) at 1 week
Statistical Analysis 2: Comparison: Prasugrel 10/10 mg; Test type: Superiority or Other; p < 0.0001, Pearson Correlation Coefficient — P-value for RPA (20 uM ADP) at 1 week
Statistical Analysis 3: Comparison: Clopidogrel 75/75 mg; Test type: Superiority or Other; p = 0.0150, Pearson Correlation Coefficient — P-value for MPA (20 uM ADP) at 1 week
Statistical Analysis 4: Comparison: Clopidogrel 75/75 mg; Test type: Superiority or Other; p = 0.0152, Pearson Correlation Coefficient — P-value for RPA (20 uM ADP) at 1 week
Statistical Analysis 5: Comparison: Prasugrel 60/10 mg; Test type: Superiority or Other; p = 0.0153, Pearson Correlation Coefficient — P-value for MPA (20 uM ADP) at 1 week
Statistical Analysis 6: Comparison: Prasugrel 60/10 mg; Test type: Superiority or Other; p = 0.0018, Pearson Correlation Coefficient — P-value for RPA (20 uM ADP) at 1 week

6. Secondary Outcome: Number of Participants With Bleeding Events by Visit According to Thrombolysis in Myocardial Infarction Study Group (TIMI) Criteria
Description: Bleeding events were classified as Major Bleeding, Minor Bleeding, or Insignificant according to TIMI criteria. Major Bleeding: any intracranial hemorrhage OR any clinically overt bleeding (including bleeding evident on imaging studies) associated with a fall in hemoglobin (Hgb) of ≥5 gm/dL from baseline. Minor Bleeding: any clinically overt bleeding (including bleeding evident on imaging studies) associated with a fall in Hgb of ≥3 gm/dL but <5 gm/dL from baseline. Insignificant Bleeding: any bleeding event that does not meet criteria for a Major or Minor Bleed.
Time Frame: End of 14 day open label (baseline); 24 Hours, 7 days, 14 days after first dose of randomized drug
Population: Safety Population - all randomized participants.
Measure: Number; unit: Participants
Arm/Group | Prasugrel 10/10 mg | Clopidogrel 75/75 mg | Prasugrel 60/10 mg
Number analyzed (Participants) | 47 | 48 | 44
Participants
  Any Bleeding at Any Time During Randomized Period | 4 | 6 | 6
  Baseline: Any Bleeding | 0 | 3 | 1
  Baseline: Insignificant Bleeding | 0 | 3 | 1
  Baseline: Minor Bleeding | 0 | 0 | 0
  Baseline: Major Bleeding | 0 | 0 | 0
  Hour 24: Any Bleeding | 0 | 0 | 1
  Hour 24: Insignificant Bleeding | 0 | 0 | 1
  Hour 24: Minor Bleeding | 0 | 0 | 0
  Hour 24: Major Bleeding | 0 | 0 | 0
  Day 7: Any Bleeding | 2 | 2 | 3
  Day 7: Insignificant Bleeding | 2 | 2 | 3
  Day 7: Minor Bleeding | 0 | 0 | 0
  Day 7: Major Bleeding | 0 | 0 | 0
  Day 14: Any Bleeding | 2 | 4 | 2
  Day 14: Insignificant Bleeding | 2 | 4 | 2
  Day 14: Minor Bleeding | 0 | 0 | 0
  Day 14: Major Bleeding | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Prasgurel 10/10 mg | Clopidogrel 75/75 mg | Prasugrel 60/10 mg
Serious Adverse Events (participants affected / at risk) | 3/47 | 0/48 | 0/44
Other Adverse Events (participants affected / at risk) | 16/47 | 25/48 | 11/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prasgurel 10/10 mg (N=47) | Clopidogrel 75/75 mg (N=48) | Prasugrel 60/10 mg (N=44)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
In-stent coronary artery restenosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prasgurel 10/10 mg (N=47) | Clopidogrel 75/75 mg (N=48) | Prasugrel 60/10 mg (N=44)
Angina pectoris (Cardiac disorders) | 1 (2) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cardiac flutter (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
Faeces hard (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0)
Exercise tolerance decreased (General disorders) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0) | 1 (1)
Feeling jittery (General disorders) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 1 (1)
Vessel puncture site haematoma (General disorders) | 0 (0) | 1 (1) | 0 (0)
Vessel puncture site reaction (General disorders) | 0 (0) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 3 (4) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 3 (4) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 4 (6) | 3 (4) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Neck injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Burning sensation (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness postural (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 4 (4) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0)
Nervousness (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Nicotine dependence (Psychiatric disorders) | 0 (0) | 1 (2) | 1 (2)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 3 (3)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1)
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyshidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (4)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Increased tendency to bruise (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 1 (2)
Haemorrhage (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
Hot flush (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days